CLINICAL TRIAL: NCT06751667
Title: Xpert Bladder Monitor: a Non-Invasive Follow-Up Tool for Detecting Relapse in High Grade or High Risk Bladder Cancer
Acronym: LIBERO
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione IRCCS Istituto Nazionale dei Tumori, Milano (Other)
Responsible Party: Principal Investigator, Nicola Nicolai, Doctor, Fondazione IRCCS Istituto Nazionale dei Tumori, Milano
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: INT 112/24
Record Dates: First submitted 2024-12-20; First posted 2024-12-30 (Actual); Last update posted 2024-12-30 (Actual); Status verified 2024-11

CONDITIONS: Bladder (Urothelial, Transitional Cell) Cancer; Bladder Cancer; Bladder Tumors; Bladder Cancer Recurrence; Cystoscopy
Keywords: Xpert Bladder Monitor; Gene Xpert
MeSH Terms: conditions — Neoplasms; Urinary Bladder Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Alternate cystoscopies and urinary biomarkers Xpert Bladder Monitor (Active Comparator): Patients with High Grade or High Risk Bladder Cancer
  Interventions: Device: Urinary biomarkers

INTERVENTIONS:
Device: Urinary biomarkers — In a bid to reduce or replace surveillance cystoscopies multiple urinary biomarkers have been evaluated for the follow-up of the bladder cancer patients. These device will reduce the number of cystoscopies

SUMMARY:
Main objectives:

Qualitative and quantitative monitoring of recurrences in patients with a previous diagnosis of high-grade bladder cancer at high risk of persistence/recurrence.

Endpoints: Presence or absence of mRNA in urine with a dichotomous result; concordance between Xpert BM and histopathological examination

Clinical relevance: reduces by half the number of (invasive) cystoscopies during follow-up. The non-invasive nature of the test could improve patient compliance with follow-up. Interventional study because it would reduce by half the number of cystoscopies during follow-up of bladder cancer which is considered the gold standard in the follow-up of this tumor. However, these markers are already CE validated and described in the European guidelines and for this reason the risk would be low.

DETAILED DESCRIPTION:
STUDY DESIGN

This prospective study is designed to assess the use of Xpert Bladder Monitor during the follow-up of patients with high grade bladder cancer. As per the guidelines, the study involves the following schedule:

* At the first outpatient check-up after diagnosis, patients will undergo cystoscopy and urinary cytology at 3 months.
* As follow-up continues, at 6 months, Xpert Bladder Monitor and 3 days urinary cytology will be performed instead of cystoscopy.
* As follow-up continues, at 9 months, standard monitoring with cistoscopy and 3 days cytology on voided urine is provided .
* As follow-up continues, at 12 months, another Xpert Bladder Monitor and 3 days urinary cytology will be performed.

The same schedule will be followed for the second year of follow-up. In the event of a positive Xpert Bladder Monitor result during follow-up, a cystoscopy will be scheduled. The study aims to enroll 50 patients for an initial follow-up of 2 years, alternating between cystoscopy and Xpert Bladder Monitor: this will involve 200 tests. The study expects to enroll patients in approximately 24 months, and with a 24-month follow-up, the study will be completed within 48 months. During the study, the possibility of extending it to a 5-year follow-up with six-monthly checks will be evaluated.The potential risk is to is not recognize a disease recurrence during follow-up at an early convenient stage. The potential benefits are related to the possibility of avoid an invasive procedure like cystoscopy which is expensive, with potential harms, surgeon-related and with a long waiting list. If patient has a positive Xpert Bladder Monitor, a cystoscopy will be performed within 30 days to verify the result.

ELEGIBILITY CRITERIA Participants will be recruited to the study only if they meet all of the inclusion criteria and none of the exclusion criteria.

4.1 Inclusion Criteria

* Age ≥ 18 years
* Has a legally acceptable representative capable of understanding the informed consent document and providing consent on the participant's behalf
* NMIBC high grade or high risk (already subjected to or currently undergoing treatment with BCG).
* No contraindications to surgery

4.2 Exclusion Criteria

* Inability or unwillingness of the participant or their legal representative to provide written informed consent
* Absolute contraindications to surgery or cystoscopy
* Patients who have previously participated in clinical protocols involving chemotherapy drugs or immunotherapy
* Patients with multiple recurrent tumors eligible for cystectomy or Muscle-Invasive Bladder Cancer (MIBC)

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Has a legally acceptable representative capable of understanding the informed consent document and providing consent on the participant's behalf
* NMIBC high grade or high risk (already subjected to or currently undergoing treatment with BCG).
* No contraindications to surgery

Exclusion Criteria:

* Inability or unwillingness of the participant or their legal representative to provide written informed consent
* Absolute contraindications to surgery or cystoscopy
* Patients who have previously participated in clinical protocols involving chemotherapy drugs or immunotherapy
* Patients with multiple recurrent tumors eligible for cystectomy or Muscle-Invasive Bladder Cancer (MIBC)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2027-01-01 (Estimated); Study Completion 2032-01-01 (Estimated)

PRIMARY OUTCOMES:
Primary objective | From enrollment to the end of treatment at 2 years
  The primary objective of this study is to qualitatively and quantitatively monitor recurrences in patients previously diagnosed with high grade or high risk bladder cancer.

SECONDARY OUTCOMES:
Secondary objective | From enrollment to the end of treatment at 2 years
  The secondary objective of the study is to verify the sensitivity, specificity and negative predictive value of miRNAs in patients with high risk bladder cancer as a laboratory tool for follow-up, to reduce an invasive test such as cystoscopy. The study also seeks to identify the ideal candidates for Xpert BM by assessing the test's specificity based on histopathological examination of cistoscopy biopsy (cold biopsy or Transurethral Resection of Bladder (TURB) samples).

IPD SHARING:
Plan to Share IPD: Undecided